CLINICAL TRIAL: NCT01212523
Title: Randomised Cross-over Pilot Study to Determine the Effects of Isoflurane and Propofol on Pulmonary Vascular Resistance in Children With Pulmonary Hypertension.
Brief Title: Effects of Propofol and Isoflurane on Pulmonary Vascular Resistance
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospitals Bristol and Weston NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Michelle White, Consultant in Paediatric Anaesthesia and Critical Care, University Hospitals Bristol and Weston NHS Foundation Trust
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: CH/2007/2476; 2009-010614-30 (Registry Identifier: EudraCT)
Record Dates: First submitted 2009-11-04; First posted 2010-09-30 (Estimated); Last update posted 2011-12-15 (Estimated); Status verified 2011-12

CONDITIONS: Hypertension, Pulmonary
Keywords: propofol; isoflurane; pulmonary hypertension; congenital heart disease
MeSH Terms: conditions — Hypertension, Pulmonary; Heart Defects, Congenital | interventions — Propofol; Isoflurane

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: propofol and isoflurane — both drugs administered at age-related dose and titrated to effect. maximum dose of propofol 15 mg/kg/hr, maximum dose of isoflurane 1.5 MAC

SUMMARY:
The investigators hypothesize that there is no difference between the effects of isoflurane and propofol anaesthesia on pulmonary vascular resistance (PVR).

ELIGIBILITY:
Inclusion Criteria:

* All children between 3 months and 16 years of age with pulmonary arterial hypertension undergoing a PVR study.

Exclusion Criteria:

* Children with a known adverse reaction to one of the study drugs eg malignant hyperpyrexia or a disorder of fatty acid oxidation.

Ages: 3 Months to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2009-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the percentage change in PVR under isoflurane anaesthesia compared with propofol anaesthesia. | 2 hours

SECONDARY OUTCOMES:
The secondary endpoints are the percentage change in mean pulomanry artery pressure (PAP), systemic vascular resistance (SVR) and mean arterial pressure (MAP). | 2 hours

CONTACTS AND LOCATIONS:
Locations (1):
- UH bristol NHS Trust, Bristol, United Kingdom